CLINICAL TRIAL: NCT00087620
Title: A Study of Capecitabine In Combination With Docetaxel vs Capecitabine Followed by Docetaxel As First-Line Treatment For Metastatic Breast Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ML17771
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: XELODA [capecitabine]

SUMMARY:
To evaluate and compare the time to progression of the combination of capecitabine (825 mg/m2 twice daily) and docetaxel (75mg/m2 i.v.) to that of capecitabine (1000 mg/m2 twice daily) until progressive disease followed sequentially by docetaxel (75 mg/m2 i.v. D1 Q3W).

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Be female and at least 18 years of age. Note: must be 19 years of age if the patient is a resident of the state of Alabama
* Be ambulatory (outpatient) and have a Karnofsky performance status of more than 70%
* Have confirmed breast cancer with locally advanced and/or metastases
* Have at least one site with defined tumor
* Have met one of the study definitions of primary or nonprimary resistance to an anthracycline-containing therapy

Exclusion Criteria:

* Pregnant/lactating women
* Women of childbearing potential with either a positive or no pregnancy test
* Women of childbearing potential unless using a reliable and appropriate contraceptive method (Postmenopausal women must have not had their period for at least 12 months to be considered of non-childbearing potential)
* Prior treatment with chemotherapy in the advanced/metastatic setting
* HER 2/neu positive status without prior treatment with trastuzumab
* Prior treatment with IV bolus 5-FU, continuous 5-FU infusion, capecitabine or other oral fluoropyrimidines
* Prior treatment with a taxane if less than 12 months passed from the time of therapy completion to relapse
* Mitomycin C or nitrosoureas within 6 weeks preceding treatment start
* Organ allografts requiring immunosuppressive therapy
* Radiotherapy to the skeleton within 4 weeks of study treatment start or insufficient recovery from the effects of prior radiotherapy
* Hormonal therapy within 10 days preceding study treatment start
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery
* Blood transfusions/growth factors to aid hematologic recovery within 2 weeks prior to study treatment start
* Participation in any investigational drug study within 4 weeks preceding treatment start
* Prior unanticipated severe reaction to fluoropyrimidine therapy
* Known hypersensitivity to 5-fluorouracil, taxanes or any of the components of capecitabine
* Requirement for concurrent use of the antiviral agent sorivudine or chemically related analogues
* Evidence of CNS metastases
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma
* Clinically significant (i.e. active) cardiac disease
* Abnormal laboratory values
* Severe renal impairment
* Serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease
* Lack of physical integrity of the upper GI tract
* Life expectancy of less than 3 months
* Unwilling/unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Little Rock, Arkansas
  - Deer Park, California
  - Greenbrae, California
  - La Jolla, California
  - Los Angeles, California
  - Orange, California
  - Aurora, Colorado
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Brooksville, Florida
  - Hollywood, Florida
  - New Port Richey, Florida
  - Augusta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Skokie, Illinois
  - Waterloo, Iowa
  - Lenexa, Kansas
  - Lafayette, Louisiana
  - Scarborough, Maine
  - Baltimore, Maryland
  - Prince Frederick, Maryland
  - Lansing, Michigan
  - Minneapolis, Minnesota
  - Reno, Nevada
  - Rochester, New York
  - Durham, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Florence, South Carolina
  - Corpus Christi, Texas
  - Richardson, Texas
  - Milwaukee, Wisconsin
  - Racine, Wisconsin